CLINICAL TRIAL: NCT00769249
Title: Correlates of Post-Traumatic Growth in Cancer Patients and Their Partners
Brief Title: Positive Changes in Quality of Life of Older Cancer Patients and Their Caregivers
Status: Withdrawn | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE8Z07; P30CA043703 (NIH); CASE8Z07 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire administration — Patients and their caregivers complete three questionnaires that will take approximately 20 minutes either by mail or telephone. The questionnaires comprise of demographic and psychosocial correlates of posttraumatic growth including age, ethnicity, socioeconomic status, education, anxiety, relationship quality, coping style, social support, and cultural beliefs about caring for elders.
Other: study of socioeconomic and demographic variables — Patients and their caregivers complete three questionnaires that will take approximately 20 minutes either by mail or telephone. The questionnaires comprise of demographic and psychosocial correlates of posttraumatic growth including age, ethnicity, socioeconomic status, education, anxiety, relationship quality, coping style, social support, and cultural beliefs about caring for elders.
Procedure: psychosocial assessment and care — Patients and their caregivers complete three questionnaires that will take approximately 20 minutes either by mail or telephone. The questionnaires comprise of demographic and psychosocial correlates of posttraumatic growth including age, ethnicity, socioeconomic status, education, anxiety, relationship quality, coping style, social support, and cultural beliefs about caring for elders.

SUMMARY:
RATIONALE: Gathering information about the positive changes in quality of life of older patients with cancer and their care givers may help doctors learn more about the disease and plan better treatment.

PURPOSE: This research study is looking at positive changes in the quality of life of older cancer patients and their caregivers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To use prior data from an existing registry (Quality of Life Survey Registry for Persons With Cancer and Family Caregivers protocol CASE-8Z05) and to expand upon these data by adding measures that capture the particularly salient concepts of the patient/caregiver dyadic relationship and posttraumatic growth.
* To identify rates and psychosocial correlates of posttraumatic growth among older adult cancer patient/spouse or partner dyads.

OUTLINE: Patients and their caregivers complete three questionnaires that will take approximately 20 minutes either by mail or telephone. The questionnaires comprise of demographic and psychosocial correlates of posttraumatic growth including age, ethnicity, socioeconomic status, education, anxiety, relationship quality, coping style, social support, and cultural beliefs about caring for elders.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient must meet the following criteria:

  * Confirmed cancer of any type
  * Currently receiving medical care at the Ireland Cancer Center at University Hospitals of Cleveland
  * Must have enrolled and participated in CASE-8Z05
* Identified available family caregiver of a patient diagnosed with stage III or IV cancer

PATIENT CHARACTERISTICS:

* Patients must meet the following criteria:

  * ECOG performance status 0-3
  * Cognitively competent to be interviewed
  * Able to speak and comprehend English
* Caregivers must be able to speak and comprehend English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Rate of posttraumatic growth | after diagnosis of cancer

CONTACTS AND LOCATIONS:
Overall Officials: T.J. McCallum, PhD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/results?term=case8z07